CLINICAL TRIAL: NCT00027235
Title: Popcorn Lung: the Discovery of a New Disease
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00036-0829
Record Dates: First submitted 2001-11-28; First posted 2001-11-29 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Lung Diseases, Interstitial; Bronchiolitis Obliterans
MeSH Terms: conditions — Lung Diseases, Interstitial; Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Recently, an epidemic of pulmonary disease has been recognized among workers in a popcorn factory in Jasper, Missouri. The exposure agent has not yet been identified, but suspects include butter flavoring and the powdered salt used in the mixing room. This disease resembles "Bronchiolitis Obliterans Syndrome", an illness that makes it difficult to breathe. Of the 117 workers studied, one year later, 25 subjects whom were working in the mixing room or in the microwave packaging area have had decreases in lung function seven times the norm for their age. Industrial hygiene experts revealed that dust concentrations of salt and other flavorings were much higher in the mixing room compared to the office and outdoor work areas. Recently, rats were exposed to vapors created by heating the butter flavor compound obtained from this plant. Six-hour exposure to vapors at very high concentration resulted in significant damage to the breathing apparatus. Thus, there is clinical, epidemiological, and animal toxicity data that appears to implicate some constituent present during the mixing of the butter flavoring, salt, and oil causing a form of obstructive airway disease that has been rapidly progressive in a number of workers. It is not clear what the pathophysiologic nature of this entity is, though it resembles Bronchiolitis Obliterans Syndrome. It is not known what the long term consequence of this will be on the active workers, nor is it clear whether preventive measures taken to reduce exposures in the mixing room and elsewhere in the plant are going to be effective.

ELIGIBILITY:
Current employees who have a decline in FEV1 larger than 200cc within the past year will be eligible to participate. All index cases will be eligible to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, Division of Pulmonary and Critical Care Medicine, St Louis, Missouri, United States